CLINICAL TRIAL: NCT06297057
Title: Acquisition and Analysis Protocol Optimization of Neurophysiological Data in Neurorehabilitation Setting: Pilot Study on Healthy Subjects
Brief Title: Acquisition and Analysis Protocol Optimization of Neurophysiological Data Neurorehabilitation Settings
Acronym: MEEGOPTI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Collaborators: University Ghent (Other); University of Padova (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021.07
Record Dates: First submitted 2024-02-08; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Healthy
Keywords: connectivity; MEEG; resting state; Mismatch Negativity (MMN); Auditory Steady State Response (ASSR)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurophysiological Recordings (Experimental): Participants suitable for hdEEG, MEG, and MUSE recordings will first undergo a neuronavigation session, and then three identical neurophysiological data acquisition sessions, one for hdEEG, one for MEG, and one for MUSE.
  The sessions will take place in three consecutive weeks, once a week, taking care that they are made at the same time of day for each participant. Finally, a structural magnetic resonance imaging (MRI) recording will be obtained for each participant.
  Each neurophysiological data acquisition session will consist of 5 blocks: 4 eyes-open and eyes-closed resting-state blocks, and one passive auditory stimulation block.
  The four blocks in the resting condition will be performed first, to avoid interference due to the passive acoustic task. The order of blocks 1 and 2, and consequently also blocks 3 and 4, representing the open-eye and closed-eye conditions will be counterbalanced between subjects and between different sessions for the same subject.
  Interventions: Other: Neurophysiological Recordings

INTERVENTIONS:
Other: Neurophysiological Recordings — Eyes-open resting-state blocks: these blocks will last 5 minutes each. Subjects will be asked to relax and not think about anything specific, keeping their eyes open and staring at a white cross in the center of a light grey screen to limit their eye movements.
  Eyes-closed resting-state blocks: these blocks will last 5 minutes each. Subjects will be asked to relax and not think about anything specific, keeping their eyes closed.
  ASSR: this block will last approximately 6 minutes. Stimuli will consist of a train of sounds presented repeatedly at high frequency.
  MMN: this block will last approximately 3 minutes. Stimuli will consist of a train of equal sounds presented alternating with a 'deviant' (rarer frequency) sound.

SUMMARY:
The study aims to optimize and validate protocols for acquiring neurophysiological data, specifically resting state functional connectivity, using advanced research techniques (hdEEG and MEG) and a user-friendly device (MUSE). Previous studies have extensively explored functional connectivity repeatability in resting conditions using functional MRI, yet few have focused on hdEEG and MEG data. Additionally, the impact of subjects' eye conditions (open or closed) during resting state recordings on network identification remains debated.

The investigation involves assessing the effect of eye conditions on brain network identification and determining the most stable and repeatable measures of functional connectivity over time. This analysis is crucial for discerning whether observed changes in patients' functional connections are intrinsic to the methodology or indicative of genuine physiological alterations.

The study aims to optimize protocols for rehabilitation by evaluating changes in functional connectivity metrics during and between experimental sessions. Furthermore, it seeks to identify the conditions (eyes closed or open) that yield more reliable and repeatable functional measurements.

Following the optimization of advanced techniques, the study explores the feasibility of utilizing the MUSE EEG system in clinical settings. MUSE, known for its portability and user-friendliness, has demonstrated quality in experimental psychology and clinical research. The objective is to establish relevant functional correspondences between measurements obtained through research techniques (hdEEG and MEG) and those acquired with MUSE.

The primary goal is to establish a protocol highlighting subjects' responses to acoustic stimuli or a reproducible pattern of resting state activity. The secondary objectives include investigating temporal and spatial characteristics of neurophysiological signals in healthy subjects over time and defining prognostic biomarkers for monitoring patients undergoing rehabilitation. This comprehensive approach aims to enhance the understanding of resting state functional connectivity and its applications in clinical settings.

Therefore, to meet these goals, the present study will consist of multiple recordings of brain activity: by high-density electroencephalography (hdEEG), magnetoencephalography (MEG), and low-density EEG with a MUSE handheld device, during five experimental blocks on healthy subjects.

DETAILED DESCRIPTION:
Participants who will be identified as suitable for hdEEG, MEG, and MUSE recording will first undergo a neuronavigation session, and then three identical neurophysiological data acquisition sessions, one for hdEEG, one for MEG, and one for MUSE.

The sessions will take place in three consecutive weeks, once a week, taking care that these recordings are made at the same time of day for each participant. Finally, a structural magnetic resonance imaging (MRI) recording will be obtained for each participant.

Each neurophysiological data acquisition session will consist of 5 blocks: 4 eyes-open and eyes-closed resting-state blocks, and one passive auditory stimulation block.

The four blocks in the resting condition will always be performed first, to avoid interference due to the passive acoustic task. The order of blocks 1 and 2, and consequently also blocks 3 and 4, representing the open-eye and closed-eye conditions will be counterbalanced between participants and between different sessions for the same participant.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65
* ability to sign an informed consent form

Exclusion Criteria:

* has suffered/is suffering from epileptic seizures.
* has had severe neurological or psychiatric disorders
* has eyesight problems that prevent him/her from reading, which she cannot correct with contact lenses (she will not be able to wear glasses during registration)
* habitually abused drugs or abused alcoholic substances
* has abused substances such as alcohol or drugs in the last three days
* is a wearer of hearing aids
* has metal and/or skull clips or other metal in any part of the head except the mouth
* has non-removable tattoos
* has piercings, earrings or other metal accessories that cannot be removed.
* is or could be pregnant (pregnancy in the first trimester)
* is a carrier of sickle cell anaemia
* is a cardiac pacemaker wearer or has an artificial heart valve
* has mechanical devices that he/she uses to administer medication
* has a surgical clip (vascular clips and metallic arterial prostheses made of ferromagnetic material)
* has a cochlear implant, a neurostimulator or a programmable hydrocephalic electrical conductor (shunt)
* has had brain surgery
* has implants or metal fragments in the body

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Neurophysiological data acquisition protocol - resting state | T1: first week, T2: second week, T3: third week
  Resting state measure from MEEG data: Power spectrum density values (delta, theta, alpha, beta, gamma frequency)
Neurophysiological data acquisition protocol - resting state | T1: first week, T2: second week, T3: third week
  Resting state measure from MEEG data: Connectivity values at source level (delta, theta, alpha, beta, gamma frequency)
Neurophysiological data acquisition protocol - auditory stimulation | T1: first week, T2: second week, T3: third week
  ASSR response (as measured from auditory stimulation)

CONTACTS AND LOCATIONS:
Locations (1):
- San Camillo IRCCS s.r.l., Venice-Lido, Venice, Italy

IPD SHARING:
Plan to Share IPD: No